CLINICAL TRIAL: NCT04945629
Title: Randomized Clinical Trial, Controlled by Conventional Treatment, of Plasma Rich in Growth Factors (PRGF®) in the Preservation of the Alveolar Ridge After Simple Molar Tooth Extractions.
Brief Title: Plasma Rich in Growth Factors in the Preservation of the Alveolar Ridge After Simple Molar Tooth Extractions.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Eduardo Anitua (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTIIMD_01_EC/20/Molares
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Dental Implantation
Keywords: exodontia; PRGF; Alveolar Ridge preservation
MeSH Terms: interventions — Blood Coagulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple suture (Active Comparator): Atraumatic exodontia followed by simple suture
  Interventions: Drug: Blood clot and simple suture
- PRGF-Endoret (Experimental): Atraumatic exodontia followed by simple suture
  Interventions: Drug: Alveolar ridge preservation with a PRP (PRGF-Endoret)

INTERVENTIONS:
Drug: Alveolar ridge preservation with a PRP (PRGF-Endoret) — Filling of the alveolus with PRGF clot and fibrin plug.
  Arms: PRGF-Endoret
Drug: Blood clot and simple suture — Filling the alveolus with blood clot
  Arms: Simple suture

SUMMARY:
This Randomized Clinical Trial aims to study the efficacy and safety of PRGF-Endoret in alveolar ridge preservation after single molar extractions. The control group is the spontaneous healing occuring after the suturing of the alveolus. The primary endpoint is the bone regeneration measured in biopsies obtained from the regenerated alveolar bone.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Clinical indication for simple tooth extraction in the posterior sectors (from the second premolar to upper and lower second molars)
* Need to place a dental implant in the same position of the extraction
* Availability of observation during the period of treatment
* Signature of the informed consent

Exclusion Criteria:

* Third molars
* Active periodontal disease
* Simultaneous extraction of two adjacent pieces in the same quadrant
* Oral dehiscence ≥ 25%
* Alveolus depth <7mm
* Loss of some wall of the alveolus
* Severe inflammation in the extraction area
* Previous diagnosis of coagulopathies
* Previous diagnosis of autoimmune disease
* Be receiving, or have received the 30 days prior to extraction treatment with radiotherapy, chemotherapy, immunosuppressants, systemic corticosteroids or anticoagulants
* Regular treatment with NSAIDs
* History of chronic hepatitis or liver cirrhosis
* Positive markers for HCV, AfHBs, HIV-I / II or TP
* Diabetes mellitus with poor metabolic control (evidence of glycated hemoglobin> 9%)
* Dialysis treatment
* Presence of malignant tumors, hemangiomas or angioma in the extraction area.
* History of ischemic heart disease in the last year
* Pregnancy or women of childbearing age who do not take action contraceptives
* Lactating women
* Previous diagnosis of metabolic bone disease
* Antiresorptive treatment
* Treatment with monoclonal antibodies
* Smoker> 10 cigarettes / day
* Any inability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Bone regeneration | 12 weeks post-extraction
  Quantity of new bone measured in bone biopsies obtained after alveolar ridge preservation

SECONDARY OUTCOMES:
Visual Analogue Score (VAS) | 3, 7 and 15 days post-extraction
  Evolution of pain assessed by the visual analog scale (VAS). Values ranging 0 to 10 (0=no pain and 10=worst pain)
Inflammation score | 3, 7 and 15 days post-extraction
  Evolution of inflammation evaluated by ordinal scale from 0 to 3 (0=no inflammation; 3=severe inflammation)
Soft tissue healing index | 3, 7 and 15 days post-extraction
  Soft tissue healing index according to the scale of Laundry. Values ranging 1 to 5 (1=poor healing, 5=excellent healing)
Changes in the dimension of the alveolar ridge | 12 weeks post-extraction
  Changes in the dimension of the alveolar ridge by means of superimposition of digital files of models of plaster after 12 weeks post-extraction
Soft tissue histomorphometric changes | 12 weeks post-extraction
  - Soft tissue histomorphometric changes after evaluated by soft tissue biopsy
Change in the bone dimensions of the alveolar ridge | 12 weeks post-extraction
  Change in the bone dimensions of the alveolar ridge evaluated by CBCT between the post-extraction day and the week 12 post-extraction.
Change in bone density | 12 weeks post-extraction
  Change in bone density (Hounsfield units) evaluated by the CBCT at three different points between the post-extraction week and 12 weeks.
Vitamin D levels | 12 weeks post-extraction
Frequency of surgical and postsurgical complications | 12 weeks post-extraction

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Eduardo Anitua, Vitoria-Gasteiz, Spain

IPD SHARING:
Plan to Share IPD: Undecided